CLINICAL TRIAL: NCT03085381
Title: A Randomized, Double-Blind and Placebo-Controlled Phase I Study to Evaluate the Safety and Primary Immunogenicity of the Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (Hansenula Polymorpha) in Chinese Female Subjects Aged 9-45 Years
Brief Title: A Phase I Study of Quadrivalent HPV Recombinant Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-HPV-1001
Record Dates: First submitted 2017-03-19; First posted 2017-03-21 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: HPV Infections
MeSH Terms: conditions — Papillomavirus Infections | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HPV vaccine (Experimental): Subjects received 3 doses of HPV vaccine according to a 0, 2, 6-month schedule.
  Interventions: Biological: HPV vaccine
- Placebo (Placebo Comparator): Subjects received 3 doses of Placebo according to a 0, 2, 6-month schedule.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: HPV vaccine
  Arms: HPV vaccine
Biological: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety and primary immunogenicity of the quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine (hansenula polymorpha) in Chinese female subjects aged 9-45 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females between, and including, 9 and 45 years of age at the time of enrolment
* Be able to provide legal identification for the sake of recruitment
* Be able to understand and sign informed consent form prior to enrollment and for subjects aged 9-17 years, they and their legal guardian(s) are supposed to understand and sign informed consent form together
* Subjects who the investigator believes that they can and will comply with the protocol requirements
* Subject must be not pregnant at the enrollment and agree to use adequate contraceptive precautions within 7 months or don't have pregnancy plan

Exclusion Criteria:

* Fever or axillary temperature> 37.0℃ before vaccination
* Previous vaccination against HPV, or planned administration/administration of a vaccine not foreseen by the study protocol within 30 days preceding first dose of vaccine; Planned to take part in other clinical research within 7 months after participating this study
* Abnormal laboratory tests parameters
* Administration of any whole blood, plasma or immunoglobulins products within 3 months preceding first vaccination
* Interval between administration of the study vaccination and any attenuated live vaccine less than 14 days, and other vaccines less than 10 days
* History of serious allergic disease requiring medical intervention (such as oral and throat swelling, difficulty breathing, hypotension or shock)
* History of to adverse event to vaccine, or allergic to some food or drug
* History of epilepsy, seizures or convulsions, or family history of mental illness
* Subjects are immunocompromised or have been diagnosed as suffering from congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis inflammation (JRA), inflammatory bowel disease or other autoimmune diseases, administration of immunosuppressants with six months prior to the first vaccine dose.
* Asplenia, functional asplenia, or any circumstances result of asplenia or splenectomy
* Subject to severe hepatorenal disease, cardiovascular disease, hypertension, diabetes, malignant tumor, all kinds of infectious diseases and acute illness, or during chronic disease acute attack period
* Medical diagnosis of coagulation abnormalities (eg, clotting factor deficiency, coagulation disorders, platelet anomaly) or obvious bruising or coagulation disorder
* During menstrual period or acute disease period of onset
* Breastfeeding, pregnancy (including pregnancy test positive), or planned to be pregnant within 7 months
* Abnormal cervical cancer screening or subject to CIN or acuteness wet wart that relevant to HPV infection in the past two years
* Planned to moveout of local before the end of the study or leave the local for a long time during the study period
* Other unsuitable factors for the study judged by investigators

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Systemic and local adverse events during the period of first dose vaccination to 30 days after last dose of vaccination | 30 days after last dose of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Zhaojun Mo, Master, Principal Investigator — Guangxi Centers for Disease Control and Prevention
Locations (1):
- Liu Zhou Centre for Disease Control and Prevention, Liuchow, Guangxi, China